CLINICAL TRIAL: NCT06367088
Title: Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Brief Title: Cadonilimab Combined With Chemotherapy as First or Second Line Treatment in Recurrent or Metastatic Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sophia
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Triple-negative Breast Cancer; Cadonilimab
Keywords: triple negative breast cancer; Cadonilimab; chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Patients were assigned to receive 10 mg/kg cadonilimab intravenously Q3W in combination with chemotherapy. The chemotherapy regimen is chosen by the physician.
  Other Names: physician's choice of chemotherapy

SUMMARY:
The prognosis of recurrent and metastatic triple negative breast cancer (TNBC) is poor, and chemotherapy is still the main treatment for TNBC. Some studies have shown that combination therapy of antibodies targeting cytotoxic T-lymphocyte antigen-4 (CTLA-4) and programmed cell death-1 (PD-1) significantly improves clinical benefit over PD-1 antibody alone. However, broad application of this combination has been limited by toxicities. Cadonilimab is a humanized immunoglobulin G1 bispecific antibody targeting PD-1 and CTLA-4. It mutates to eliminate Fc receptor and complement-mediated cytotoxic effects. The purpose of this study is to evaluate the efficacy and safety of Cadonilimab combined with chemotherapy as a first or second-line treatment of recurrent and metastatic TNBC. This study is a multicenter, single arm, phase II, non randomized, open label, Simon two-stage design. It is planned to enroll 27 late stage TNBC patients.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic TNBC patients;
* TNBC defined by immunohistochemistry as ER<1%, PR<1%, Her2=0~1+, or 2+ while HER2 Fish test shows no amplification；
* Previous received no or only first line chemotherapy treatment for recurrent or metastatic TNBC；When the time between cancer metastasis and the end of adjuvant chemotherapy exceeds 1 year, the systemic chemotherapy for metastasis treatment is recorded as first-line treatment; When less than 1year, the systemic chemotherapy for metastasis treatment is recorded as second-line treatment；
* ages 18 to 75 years at the time of signing the informed consent form (ICF);
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
* expected survival of ≥3 months; at least one measurable lesion per RECIST (version1.1);
* acceptable renal and liver function;

Exclusion Criteria:

* They had received ICIs (i.e., anti-PD-1 antibodies, anti-PD-L1 antibodies, and anti-CTLA-4 antibodies.)；
* Patients with active central nervous system (CNS) metastatic lesions or meningeal metastases；
* Patients with an active autoimmune disease that requires systemic treatment in the past two years；
* A known history of primary immunodeficiency；
* Pregnant or lactating women；
* Previous or current abnormalities of any disease, treatment, laboratory tests may confuse the study results, affect the subject's participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
AE | From the time of informed consent signed through 90 days after the last dose of drug
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

OTHER OUTCOMES:
Progression-free survival | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK104 until death due to any cause.
Disease control rate | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Zhao, PhD, Study Chair — Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No